CLINICAL TRIAL: NCT01688544
Title: Phase 1 Study to Evaluate the Effect of CYP Polymorphism and Gender on the Pharmacokinetics and Pharmacodynamics of Ilaprazole After Multiple Dosing
Brief Title: Pharmacokinetic/Pharmacodynamic Study of Ilaprazole to Evaluate the Effect of CYP Genetic Polymorphism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-112
Record Dates: First submitted 2011-12-06; First posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Ilaprazole; Intragastric pH; Serum Gastrin; Pharmacokinetics
MeSH Terms: interventions — ilaprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ilaprazole (Experimental): Before Ilaprazole dosing, 24 hours intragastric pH monitoring is performed as baseline value.
  After 7 days dosing of Ilaprazole 10 mg, 24 hours intragastric pH monitoring, serum gastrin level check, and pharmacokinetic sampling is performed
  Interventions: Drug: Ilaprazole

INTERVENTIONS:
Drug: Ilaprazole — Ilaprazole 10 mg for 7 days
  Other Names: 2-[(4methoxy-3-methyl)-2-pyridinyl] methylsulfinyl-; 5-(1H-pyrrol-1yl)-1H-benzimidazole

SUMMARY:
Ilaprazole is a novel proton pump inhibitor and metabolized by CYP3A4 and 2C19. Thus genetic polymorphisms of CYP3A4 and 2C19 may have effect on the pharmacokinetics and pharmacodynamics of Ilaprazole.

DETAILED DESCRIPTION:
Effects of genetic polymorphisms on the pharmacokinetics or pharmacodynamics were measured in healthy Korean volunteers

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteer between 20 and 45 years of age and within 20% of ideal body weight
* No congenital or acquired chronic disease
* appropriate for the study judging from examinations (hematology, chemistry, urinalysis and so on), vital sign and ECG results
* sign the informed consent form prior to study participation

Exclusion Criteria:

* received any metabolizing enzymes or transporters inducing or inhibiting drugs like barbiturates within 1 month prior to the date of first drug administration
* history of hypersensitivity against drugs or clinically significant allergic diseases
* abnormal laboratory results
* positive result for helicobacter pylori infection from the Urea Breath Test
* alcohol or drug abuser
* pregnant or lactating
* donated whole blood within 60days prior to the study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
24 hour intragastric ph | After 7 days dosing of Ilaprazole 10 mg

SECONDARY OUTCOMES:
Pharmacokinetic parameters (Cmax, AUC) of Ilaprazole and its metabolite | After 7 days dosing of Ilaprazole
Serum Gastrin level | After 7 days dosing of Ilaprazole

CONTACTS AND LOCATIONS:
Overall Officials: JaeGook Shin, MD,PhD, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hoapital Clinical Trial Center, Busan, Busan, South Korea